CLINICAL TRIAL: NCT01382290
Title: Magnetic Resonance Imaging of the Spine
Acronym: MRIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were enrolled, due to logistic difficulties, no funding was acquired.
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Richard Jones, PhD, Children's Healthcare of Atlanta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI DIffusion Spine
Record Dates: First submitted 2005-09-13; First posted 2011-06-27 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Tethered Cord; Chiari I Malformation
Keywords: MRI; Spine; Diffusion
MeSH Terms: conditions — Spinal Cord Injuries; Arnold-Chiari Malformation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MRI

SUMMARY:
Diffusion-weighted (DW) magnetic resonance imaging (MRI) imaging is a well established method for detecting acute injury to the brain and is used on all children undergoing an MRI brain scan at Children's Healthcare of Atlanta. The possibility of using DW MRI to study other areas of the body, such as the spinal cord, has been recognised as having great clinical potential. However, two main problems have hindered the clinical application of the technique; firstly, the extreme motion sensitivity of the technique meant that respiratory motion have hampered clinical studies. Secondly, the close proximity of the spinal cord to the bones in the spinal column complicates the application of the techniques developed for the brain to the spine. Recently, several techniques have been developed which address these problems and these are now available on the MRI scanners used at Children's Healthcare of Atlanta.

We now wish to evaluate how well these techniques work on children in a routine clinical setting. For this reason we wish to add a single scan of the spine to the imaging protocol of children receiving a routine scan of the brain or spine. This will permit us to evaluate the image quality in both normal and abnormal spines. We plan on enrolling 60 patients with normal spines and 30 patients with abnormal spines. No additional sedation and/or contrast will be required and the additional imaging time for the diffusion studies will be less than 10 minutes. Parental consent will be a pre-requisite for any patient to be enrolled into the study.

DETAILED DESCRIPTION:
Background and significance

Diffusion-weighted (DW) magnetic resonance imaging (MRI) imaging is a well established method for detecting acute ischaemic injury in the brain and is being increasingly applied to the study of brain structure and organisation (1,2). The technique provides information on the motion of water molecules and uses no ionising radiation. The possibility of using DW MRI to probe neuronal microstructures in highly ordered neuronal systems, such as the spinal cord, has been recognised as having great clinical potential. However, the combination of susceptibility artefacts from the surrounding bony structures, motion of the cerebrospinal fluid (CSF), carotid and vertebral artery pulsations and respiratory motion have hampered clinical studies. Recently, several techniques have been developed to address these problems (3,4) and two of these methods will shortly be available for use at the Scottish Rite campus of CHOA.

We propose to apply DW imaging of the spine to the following groups of patients :

1. Patients with tethered cords.
2. Patients with Chiari I malformations.
3. Normal children undergoing a MRI of the spine.

All of the studies would be performed on children who have already been referred for a MRI and the diffusion sequences would be performed after the requested MRI exam is complete. No additional sedation and/or contrast would be required. Informed consent would be requested from the parents for all of these studies. The additional imaging time required for the diffusion studies would be less than 10 minutes. We plan on enrolling 60 patients with normal spines and 30 patients with abnormal spines in this study.

Tethered cord. Tethered spinal cords are a group of complex developmental malformations of the spinal cord of which the most common cause is children with repaired spina-bifida or myelomeningocele. Although these are usually operated on shortly after birth, all repaired myelomeningoceles have some degree of tethering. The basic problem is exacerbated because as children grow their spinal cords do not grow as quickly as their spinal columns, so the spinal cord must be able to freely ascend on the inside of the spinal column during growth. If various abnormal structures are holding onto the spinal cord from below it stretches the spinal cord, leading to chronic local ischaemia, which can in turn lead to a progressive loss of function. The signs and symptoms associated with cord tethering are often non-specific and are poorly understood. Diffusion MRI may be very useful in the monitoring of tethered cords since initial studies on adults with cervical spondylosis have implied that it is more sensitive than conventional MRI imaging in depicting pathological changes within the spinal cord. Hence diffusion MRI has the potential to be a more sensitive method of determining if the cord is under stress due to tethering and hence in need of surgery.

Chiari I malformation A Chiari I malformation is a condition characterised by an abnormal inferior projection of the cerebellar tonsils through the foramen magnum, into the upper cervical spinal canal. If the degree of projection is small then the condition is generally referred to as tonsilar ectopia. Chiari I malformations may be associated with other anomalies, most commonly hydrosyringomyelia (which in turn can lead to neurologic deficits and scoliosis) and hydrocephalus. Symptoms of a Chiari I malformation most often begin during infancy, although they may be delayed until adolescence or adulthood. Symptoms are often non-specific and usually include headache, vomiting, muscle weakness in the head and face, difficulty swallowing, and varying degrees of mental impairment. Paresis or paralysis of the arms and legs may also occur. As they grow older, adolescents and adults with Chiari I malformation who previously were asymptomatic may show signs of progressive brain impairment, such as involuntary, rapid, downward eye movements. The pathophysiology of syrinx development (hydrosyringomyelia) is understood to be a state of chronic interstitial edema of the spinal cord due to an accumulation of extracellular fluid.

A diagnosis of Chiari I malformation is generally made using a conventional MRI scan and is often an incidental finding during an evaluation of other abnormalities, making an interpretation of the significance of the imaging findings difficult. Patients that have symptoms which potentially indicate abnormally positioned tonsils can have normal imaging findings, tonsilar ectopia or mild Chiari I malformation. In the case that the cerebellar tonsils are not clearly abnormal, according to our conventional imaging diagnostic criteria, it can be difficult to determine the cause of the symptoms. They may be caused by the low tonsils, in which case a surgical decompression would be performed, or they may simply be incidental findings.

A further problem in determining a strategy for managing patients with a Chiari I malformation is that the criteria for surgical intervention are nebulous. Some patients are symptomatic with only a minor degree of tonsillar ectopia and others with severe displacement of the cerebellar tonsils into the upper spinal canal have no symptoms. Since the correction of a Chiari I malformation requires surgery it is generally reserved for patients showing clear evidence of progressive clinical symptoms. Any technique that can provide information on pathological changes within the spinal cord would be a very important complement to the clinical data and the anatomical information provided by conventional MRI. At present it is difficult to predict which patients are predisposed to developing syringomyelia on the basis of conventional imaging findings alone and DW-MRI may be able to provide useful complementary information.

Normal patients. To date the only information regarding the values for diffusion within the spinal cord comes from a limited number of studies on normal, adult, volunteers. It is known that the diffusion properties of the brain vary significantly with age and it is expected that the diffusion properties of the spine will show a similar variation. Thus, in order to be able to properly interpret the results of the studies on children with suspected pathology it is necessary to have a control group in order to allow normal values for different age ranges to be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tethered cords.
* Patients with Chiari I malformations.
* Normal children undergoing a MRI of the spine.

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jones, PhD, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (1):
- Childrens Healthcare at Scottish Rite, Atlanta, Georgia, United States